CLINICAL TRIAL: NCT01431456
Title: A Randomized Pilot Study Comparing the Safety of DAbigatran and RIvaroxaban Versus NAdroparin in the Prevention of Venous Thromboembolism After Knee Arthroplasty Surgery
Brief Title: Safety of DAbigatran and RIvaroxaban Versus NAdroparin in the Prevention of Venous Thromboembolism After Knee Arthroplasty Surgery
Acronym: DARINA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Martini Hospital Groningen (Other)
Responsible Party: Principal Investigator, Marinus van Hulst, Hospital Pharmacist, Martini Hospital Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DARINA
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Venous Thromboembolism
Keywords: Prevention; venous thromboembolism after knee arthroplasty
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran; Rivaroxaban; Nadroparin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dabigatran (Active Comparator): Dabigatran
  Interventions: Drug: Dabigatran
- Rivaroxaban (Active Comparator): Rivaroxaban
  Interventions: Drug: Rivaroxaban
- Nadroparin (Active Comparator): Nadroparin
  Interventions: Drug: Nadroparin

INTERVENTIONS:
Drug: Dabigatran — Dabigatran
  Arms: Dabigatran
Drug: Rivaroxaban — Rivaroxaban
  Arms: Rivaroxaban
Drug: Nadroparin — Nadroparin
  Arms: Nadroparin

SUMMARY:
Rationale:

After total knee arthroplasty (TKA) surgery, patients are at risk to develop venous thromboembolism (VTE) or deep venous thrombosis (DVT) potentially resulting in a fatal pulmonary embolism (PE). Two novel agents, dabigatran and rivaroxaban, recently gained market authorisation for prevention of venous thromboembolism after knee arthroplasty.

However, there are no clinical trials with dabigatran and/or rivaroxaban and the comparator nadroparin.

Nadroparin is used in the most Dutch departments of orthopaedic surgery after total knee arthroplasty. Also safety of the new oral agents with long term use of 42 days is not available for total knee arthroplasty.

Our aim is to compare the long term use of dabigatran and rivaroxaban versus nadroparin on safety after total knee arthroplasty (TKA) in a clinical explorative pilot study by observing the incidence of major bleeding and clinical relevant non-major bleeding using a standardized model of bleeding definitions.

Objective:

The primary objective of this study is to compare the clinical safety with long term use of the oral once daily unmonitored thrombin inhibitors dabigatran and rivaroxaban versus subcutaneous administered nadroparin by observing the incidence of major bleeding and clinical relevant non-major bleeding in patients after knee arthroplasty surgery.

The secondary objectives of this study are effectivity of the agents, compliance, hospital stay, re-hospitalisation, outpatient clinic visits and interventions following complications. Additionally, coagulation monitoring, knee flexion range of motion, Knee injury and Osteoarthritis Outcome Score (KOOS), Knee Society Score (KSS) and relationship between health statuses and surgery parameters will be evaluated.

Study design:

The study is designed as non-inferiority randomized open label controlled pilot study. A total of 150 patients will be included, 50 patients in each treatment group (dabigatran, rivaroxaban and nadroparin).

Study population:

Patients ≥ 18 years and weighing more than 40 kg, participate in the 'joint care program' for primary elective total knee arthroplasty and want to provide signed informed consent are eligible for the study.

Intervention:

Patients receive subcutaneously nadroparin or oral rivaroxaban or oral dabigatran after knee replacement surgery.

Main study parameters/endpoints:

The primary safety outcome is the incidence of bleeding events occurring during the study period of 135 days (including follow-up). Major bleeding events and clinically relevant non-major bleeding events were defined according to accepted guidelines.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years and weighing more than 40 kg who are scheduled for primary elective total knee arthroplasty according to the 'joint care program' and want to provided signed informed consent are eligible for the study.

Exclusion Criteria:

* a known inherited or acquired clinically significant active high risk of bleeding or bleeding disorder;
* major surgery, trauma, uncontrolled severe arterial hypertension, or myocardial infarction within the last 3 months;
* history of acute intracranial disease or hemorrhagic stroke;
* gastrointestinal or urogenital bleeding or ulcer disease within the last 6 months;
* cirrhotic patients with moderate hepatic impairment (aspartate or alanine aminotransferase (AST, ALT) levels higher than 2x the upper limit of the normal range (ULN) within the last month);
* severe renal insufficiency (creatinine clearance < 30 mL/min);
* treatment with anticoagulants during study drug treatment;
* active malignant disease;
* pregnancy or breastfeeding;
* and unable to give informed consent.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The primary safety outcome is the incidence of bleeding events occurring during the study period of 135 days (including follow-up). Major bleeding events and clinically relevant non-major bleeding events were defined according to accepted guidelines | 135 days
  Major and clinically relevant non-major bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Martini Ziekenhuis, Groningen, Netherlands

REFERENCES:
- [Derived] van der Veen L, Segers M, van Raay JJ, Gerritsma-Bleeker CL, Brouwer RW, Veeger NJ, van Hulst M. Bleeding complications of thromboprophylaxis with dabigatran, nadroparin or rivaroxaban for 6 weeks after total knee arthroplasty surgery: a randomised pilot study. BMJ Open. 2021 Jan 18;11(1):e040336. doi: 10.1136/bmjopen-2020-040336. PMID 33462096
- [Derived] Veen Lv, van Raay JJ, Gerritsma-Bleeker CL, Veeger NJ, Hulst Mv. Direct treatment comparison of DAbigatran and RIvaroxaban versus NAdroparin in the prevention of venous thromboembolism after total knee arthroplasty surgery: design of a randomised pilot study (DARINA). BMJ Open. 2013 Jan 24;3(1):e002218. doi: 10.1136/bmjopen-2012-002218. PMID 23355673